CLINICAL TRIAL: NCT03779919
Title: The Therapeutic Effect of the Extracorporeal Shock Wave Therapy on Shoulder Calcific Tendinitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chimei Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMMC10709-004
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Calcific Tendinitis
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Energy (Experimental): Extracorporeal shock wave therapy with 0.3 millijoule/mm2 of 3000 shots will be administered via sonographic guidance of the target calcific tendinitis.
  Interventions: Device: extracorporeal shock wave
- Low Energy (Experimental): Extracorporeal shock wave therapy with 0.05 millijoule/mm2 of 3000 shots will be administered via sonographic guidance of the target calcific tendinitis.
  Interventions: Device: extracorporeal shock wave
- Sham (Placebo Comparator): Extracorporeal shock wave therapy with 0 millijoule/mm2 of 3000 shots will be administered via sonographic guidance of the target calcific tendinitis.
  Interventions: Device: extracorporeal shock wave

INTERVENTIONS:
Device: extracorporeal shock wave — Extracorporeal shock wave therapy uses acoustic waves to fragment calcific deposits. Variables of the settings include dose (low or high energy), duration (impulses), and the interval of administration.

SUMMARY:
Calcific tendinopathy of the shoulder is often self-limited with a relatively benign clinical course. Therefore, first-line therapy should be conservative and focused on symptom relief. However, studies show patients with Large volume deposits (e.g. ≥1500 mm3) and Subacromial extension of the deposits respond poorly to initial treatment such as analgesic medication, glucocorticoid injection, and physical therapy. For those refractory cases, extracorporeal shock wave therapy is introduced and shows resolution of symptoms and improvement in shoulder function in approximately 70 percent of patients.

Extracorporeal shock wave therapy uses acoustic waves to fragment calcific deposits. Variables of the settings include dose (low or high energy), duration (impulses), and the interval of administration. However, an optimum value for the total cumulative dose of energy that should be administered has not yet been defined. Our study thus aim to find out the dosage effect of ESWT on the calcific debris sizes, pain, daily living functions, and shoulder range of motions in the calcific tendinitis patients.

DETAILED DESCRIPTION:
Calcific tendinopathy of the shoulder is caused by unknown etiology characterized by the formation of calcific deposits in on or several tendons of the rotator cuff muscles: supraspinatus, infraspinatus, teres minor, and subscapularis muscles. The calcific deposits is often composed of poorly crystallized hydroxyapatite, an inorganic component of bone tissue, but the pathogenesis of rotator cuff disorders is still incomplete.

The clinical presentations of calcific tendinopathy typically involve shoulder pain similar to that experienced by patients with rotator cuff tendinopathy or shoulder impingement syndrome. Pain is the cardinal symptom and is localized on the top or lateral aspect of the shoulder or both, often with radiation towards the insertion of the deltoid. The onset of pain is gradual and unassociated with trauma. Daily activities involving overhead motions, such as putting on a shirt or brushing hair, can be painful, thus decreasing quality of life immensely.

Calcific tendinopathy of the shoulder is often self-limited with a relatively benign clinical course. Therefore, first-line therapy should be conservative and focused on symptom relief. However, some remain ineffective to the initial treatment. For those refractory cases, extracorporeal shock wave therapy (ESWT) is introduced and shows resolution of symptoms and improvement in shoulder function in approximately 70 percent of patients.

ESWT uses acoustic waves to fragment calcific deposits. Variables of the settings include dose (low or high energy), duration (impulses), and the interval of administration. However, an optimum value for the total cumulative dose of energy that should be administered has not yet been defined. Our study thus aim to find out the dosage effect of ESWT on the calcific debris sizes, pain, daily living functions, and shoulder range of motions in the calcific tendinitis patients.

The study will be a prospective assessor-blinded randomized controlled trial. Patients who have calcific tendinitis diagnosed by shoulder sonography or X-ray, fail to improve despite appropriate conservative treatment for three months will be recruited. The subjects will be randomized distributed in 3 groups: High Energy, Low Energy, and Sham groups, and each group has 30 patients.

Upon completion of the study, the result will show whether different dosage of ESWT has different therapeutic effects on shoulder calcific tendinitis. In the future, the study may be the foundation of the ESWT treatment guideline for rotator calcific tendinitis.

ELIGIBILITY:
Inclusion Criteria:

．age 20-70 with calcific tendinitis via sonography or x-ray in rotator cuff

Exclusion Criteria:

．no shoulder fracture, no abnormality, gout or autoimmune disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-11-18 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
changes from baseline in the calcium deposits | one month and 3 months after shock wave
  Calcium deposits will be measured via X-ray or sonography.

SECONDARY OUTCOMES:
functional score | one month and 3 months after shock wave
  The 100-point Constant score will be used to provide an overall clinical assessment of the shoulder with respect to the degree of pain, the patient's ability to perform normal tasks of daily living (maximal score, 35), and the active range of motion and power of the shoulder, or torque (maximal score, 65)
pain score | one month and 3 months after shock wave
  The severity of pain at night and during the day, both on movement and at rest, is assessed by means of a visual-analogue scale that ranges from 0 (no pain) to 10 (severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Han Cheng, MD, Principal Investigator — ChiMei Medical Center, Taiwan, R.O.C.
Locations (1):
- ChiMei Medical Center, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No